CLINICAL TRIAL: NCT04047706
Title: Combination of Checkpoint Inhibition and IDO1 Inhibition Together With Standard Radiotherapy or Chemoradiotherapy in Newly Diagnosed Glioblastoma. A Phase 1 Clinical and Translational Trial
Brief Title: Nivolumab, BMS-986205, and Radiation Therapy With or Without Temozolomide in Treating Patients With Newly Diagnosed Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU 18C02; NCI-2019-04922 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00209583; NU 18C02 (Other: Northwestern University); P30CA060553 (NIH); P50CA221747 (NIH)
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — linrodostat; Nivolumab; Radiotherapy; Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Methylated Cohort (radiation, temozolomide, BMS-986205 25mg QD, nivolumab) (Experimental): RADIATION THERAPY: Patients with MGMT methylated promoter undergo radiation therapy 5 days per week (Monday-Friday) for up to 6 weeks. Patients also receive temozolomide PO QD, IDO1 inhibitor BMS-986205 PO QD, and nivolumab IV over 30 minutes every 2 weeks for up to 6 weeks in the absence of disease progression, unacceptable toxicity, withdrawal of consent, the study ends, or until Q4W dosing begins.
  MAINTENANCE THERAPY: Patients receive IDO1 inhibitor BMS-986205 PO QD on days 1-28 and nivolumab IV over 30 minutes on days 1 and 15 of cycles 1-5 and on day 1 of subsequent cycles. Within 4 weeks of radiation therapy completion, patients also receive temozolomide PO QD on days 1-5 of cycles 2-6. Cycles repeats every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: IDO1 Inhibitor BMS-986205 25mg; Drug: Nivolumab; Radiation: Radiation Therapy; Drug: Temozolomide
- Unmethylated Cohort (radiation, BMS-986205 50mg QD, nivolumab) (Experimental): RADIATION THERAPY: Patients with MGMT unmethylated promoter undergo radiation therapy 5 days per week (Monday-Friday) for up to 6 weeks. Patients also receive IDO1 inhibitor BMS-986205 PO QD and nivolumab IV over 30 minutes every 2 weeks for up to 6 weeks in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive IDO1 inhibitor BMS-986205 PO QD on days 1-28 and nivolumab IV over 30 minutes on days 1 and 15 of cycles 1-5 and on day 1 of subsequent cycles. Cycles repeats every 28 days for up to 2 years in the absence of disease progression, unacceptable toxicity, withdrawal of consent, the study ends, or until Q4W dosing begins.
  Interventions: Drug: Nivolumab; Radiation: Radiation Therapy; Drug: IDO1 Inhibitor BMS-986205 50 mg
- Unmethylated Cohort (radiation, BMS-986205 100mg QD, nivolumab) (Experimental): RADIATION THERAPY: Patients with MGMT unmethylated promoter undergo radiation therapy 5 days per week (Monday-Friday) for up to 6 weeks. Patients also receive IDO1 inhibitor BMS-986205 PO QD and nivolumab IV over 30 minutes every 2 weeks for up to 6 weeks in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive IDO1 inhibitor BMS-986205 PO QD on days 1-28 and nivolumab IV over 30 minutes on days 1 and 15 of cycles 1-5 and on day 1 of subsequent cycles. Cycles repeats every 28 days for up to 2 years in the absence of disease progression, unacceptable toxicity, withdrawal of consent, the study ends, or until Q4W dosing begins.
  Interventions: Drug: Nivolumab; Radiation: Radiation Therapy; Drug: IDO1 Inhibitor BMS-986205 100 mg

INTERVENTIONS:
Drug: IDO1 Inhibitor BMS-986205 25mg — Given PO
  Other Names: BMS 986205; BMS-986205; BMS986205; IDO-1 Inhibitor BMS-986205; Indoleamine-pyrrole 2,3-Dioxygenase Inhibitor BMS-986205; ONO-7701
  Arms: Methylated Cohort (radiation, temozolomide, BMS-986205 25mg QD, nivolumab)
Drug: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ
  Arms: Methylated Cohort (radiation, temozolomide, BMS-986205 25mg QD, nivolumab)
Drug: IDO1 Inhibitor BMS-986205 50 mg — Given PO
  Other Names: BMS 986205; BMS-986205; BMS986205; IDO-1 Inhibitor BMS-986205; Indoleamine-pyrrole 2,3-Dioxygenase Inhibitor BMS-986205; ONO-7701
  Arms: Unmethylated Cohort (radiation, BMS-986205 50mg QD, nivolumab)
Drug: IDO1 Inhibitor BMS-986205 100 mg — Given PO
  Other Names: BMS 986205; BMS-986205; BMS986205; IDO-1 Inhibitor BMS-986205; Indoleamine-pyrrole 2,3-Dioxygenase Inhibitor BMS-986205; ONO-7701
  Arms: Unmethylated Cohort (radiation, BMS-986205 100mg QD, nivolumab)

SUMMARY:
This phase I trial studies the side effects of nivolumab, BMS-986205, and standard radiation therapy with or without temozolomide in treating patients with new diagnosed glioblastoma. Immunotherapy with nivolumab, may induce changes in body?s immune system and may interfere with the ability of tumor cells to grow and spread. BMS-986205 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving nivolumab and BMS-986205 may work better compared to radiation therapy and temozolomide alone in treating patients with newly diagnosed glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of nivolumab in combination with IDO1 inhibitor BMS-986205 (BMS986205) and radiation in newly diagnosed MGMT promoter unmethylated glioblastoma and MGMT promoter methylated glioblastoma.

SECONDARY OBJECTIVES:

I. Descriptive survival analyses (overall survival [OS] and OS at 12 months [OS12]) in patients with MGMT unmethylated and MGMT methylated promoter.

II. Progression free survival (PFS) and PFS at 6 months (PFS6) in patients with MGMT unmethylated and MGMT methylated promoter.

III. Radiographic response rates (RR) as determined by Response Assessment in Neuro-Oncology (RANO) and immunotherapy (i)RANO criteria in patients with MGMT unmethylated and MGMT methylated promoter.

EXPLORATORY OBJECTIVES:

I. Determine the T-cell changes that occur in glioblastoma (GBM) treated with nivolumab in combination with BMS-986205 and radiation.

II. Correlate T-cell changes and IDO1 expression with patient outcomes.

OUTLINE: This is a dose-escalation study of IDO1 inhibitor BMS-986205. Patients are assigned to 1 of 2 cohorts.

COHORT I:

RADIATION THERAPY: Patients with MGMT methylated promoter undergo radiation therapy 5 days per week (Monday-Friday) for up to 6 weeks. Patients also receive temozolomide orally (PO) once daily (QD), IDO1 inhibitor BMS-986205 PO QD, and nivolumab intravenously (IV) over 30 minutes every 2 weeks for up to 6 weeks in the absence of disease progression, unacceptable toxicity, withdrawal of consent, the study ends, or until Q4W dosing begins.

MAINTENANCE THERAPY: Patients receive IDO1 inhibitor BMS-986205 PO QD on days 1-28 and nivolumab IV over 30 minutes on days 1 and 15 of cycles 1-5 and on day 1 of subsequent cycles. Within 4 weeks of radiation therapy completion, patients also receive temozolomide PO QD on days 1-5 of cycles 2-6. Cycles repeats every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

COHORT II:

RADIATION THERAPY: Patients with MGMT unmethylated promoter undergo radiation therapy 5 days per week (Monday-Friday) for up to 6 weeks. Patients also receive IDO1 inhibitor BMS-986205 PO QD and nivolumab IV over 30 minutes every 2 weeks for up to 6 weeks in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive IDO1 inhibitor BMS-986205 PO QD on days 1-28 and nivolumab IV over 30 minutes on days 1 and 15 of cycles 1-5 and on day 1 of subsequent cycles. Cycles repeats every 28 days for up to 2 years in the absence of disease progression, unacceptable toxicity, withdrawal of consent, the study ends, or until Q4W dosing begins.

After completion of study treatment, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a newly diagnosed histologically confirmed diagnosis of any grade IV glioma with documentation of MGMT methylation status. The histological diagnosis can be obtained either from a brain biopsy or from a neurosurgical resection of the tumor

  * Note: Study enrollment is to be within 5 weeks from diagnostic surgery or biopsy
  * Note: Pyrosequencing to determine MGMT methylation status will be performed at Northwestern Memorial Hospital as standard of care (SOC)
* Tumor tissue specimens from the GBM surgery or biopsy for central pathology review and exploratory analysis of immunocorrelative studies, if available (no minimum requirement)
* For subjects who had undergone tumor resection, preoperative gadolinium (Gd)-magnetic resonance imaging (MRI) and immediate postoperative Gd-MRI performed within < 72 hours after surgery or biopsy is recommended. If computed tomography (CT) scans were performed perioperatively, an MRI should be performed before initiation of study treatment
* Patients must exhibit a Karnofsky performance score of >= 70%
* Stable or decreasing dose of steroids for >= 7 days prior to registration

  * Note: Patients must be off of all steroids at the time of initiation of study treatment (day 1 [D#1])
* Patients must have adequate organ and bone marrow function at registration, as defined below:
* Absolute neutrophil count >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Creatinine or creatinine clearance =<1.5 times upper limit of normal or >= 60 mL/min
* Hemoglobin >=10 mg/dL

  * Blood transfusion allowed
* Total bilirubin =< 1.5 times upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SPGT]) =< 2.5 times above upper limit of normal
* Alkaline phosphatase =< 2.5 times above upper limit of normal
* Females of child-bearing potential (FOCBP) and males must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 5 months following completion of therapy. Should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Due to the potential interaction with study drug(s), contraceptions that use hormones are not considered to be highly effective for FOCBP participants in this study.

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy. Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* Males who are sexually active with FOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatment plus 7 months after the last dose of the study treatment (i.e., 90 days [duration of sperm turnover] plus the time required for nivolumab to undergo approximately 5 half-lives). In addition, male participants must be willing to refrain from sperm donation during this time. Male participants with partners who are FOCBP are required to use a condom for study duration and until end of relevant systemic exposure defined as 7 months after the end of study treatment. This criteria applies to azoospermic males as well
* FOCBP must have a negative serum pregnancy test within 14 days of registration on study and within 24 hours of beginning study treatment
* Clinically normal cardiac function without history of ischemic heart disease in the past 6 months and normal 12 lead electrocardiogram (ECG)
* Patients must have recovered from the effects of surgery, postoperative infection, and other complications before study registration
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients who have had chemotherapy within 2 years prior to entering the study are not eligible
* Patients who have received brain radiation therapy (RT) are not eligible
* Patients may not be receiving any other investigational agents. Patients may not have received an investigational agent within the past 30 days prior to the initiation of study treatment
* Patients with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications are not eligible

  * Note: Inhaled or topical steroids, and adrenal replacement steroid doses >= 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Patients with an active, known or suspected autoimmune disease are not eligible. Patients with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Participants with a personal or family (i.e., in a first-degree relative) history or presence of cytochrome b5 reductase deficiency (previously called methemoglobin reductase deficiency) or other diseases that puts them at risk of methemoglobinemia are not eligible. All participants will be screened for methemoglobin levels prior to registration
* Participants with a history of G6PD deficiency or other congenital or autoimmune hemolytic disorders are not eligible. All participants will be screened for G6PD levels prior to registration
* Participants with active interstitial lung disease (ILD)/pneumonitis or with a history of ILD/pneumonitis requiring steroids are not eligible
* Patients with a history of recent prior malignancy are not eligible. Subjects with curatively treated cervical carcinoma in situ or non-melanoma basal cell carcinoma of the skin, or subjects who have been free of other malignancies for >= 2 years are eligible for this study
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab, temozolomide or BMS-986205 are not eligible
* Patients who have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways are not eligible
* Patients who have had prior treatment with BMS-986205 or any other IDO1 inhibitors are not eligible
* Patients who have received treatment with botanical preparations (e.g., herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 14 days prior to registration are not eligible
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Hypertension that is not controlled on medication
  * Ongoing or active infection requiring systemic treatment
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient?s safety or study endpoints
* Female patients who are pregnant or nursing are not eligible
* Patients who have quantitative or qualitative G6PD assay results suggesting underlying G6PD deficiency are not eligible
* Patients who have blood methemoglobin > upper limit of normal (ULN), assessed in an arterial or venous blood sample or by co-oximetry are not eligible
* Patients with a concurrent illness, including severe infection, which may jeopardize the ability of the subject to receive the procedures outlined in this protocol with reasonable safety are not eligible. Concomitant use of strong inhibitors of CYP3A4/1A2 within 1 week or 5 half-lives (whichever is longer) or strong inducers of CYP3A4/1A2 within 2 weeks or 5 halflives (whichever is longer) is not permitted
* Patients with a placement of Gliadel wafer at surgery are not eligible
* Patients receiving Optune therapy are not eligible
* Patients who are unable to undergo Gd-MRI are not eligible
* Patients with current known alcohol dependence or drug abuse are not eligible
* Patients with a history or presence of hypersensitivity or idiosyncratic reaction to methylene blue are not eligible
* Patients with a prior history of serotonin syndrome are not eligible
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).

  * Note: Testing for HIV must be performed at sites where mandated locally
* Patients who have any positive test result for hepatitis B virus or hepatitis C virus indicating presence of virus, e.g., hepatitis B surface antigen (HBsAg, Australia antigen) positive, or hepatitis C antibody (anti-HCV) positive (except if hepatitis c virus [HCV] ribonucleic acid [RNA] negative) are not eligible
* Patients with the presence of any familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule are not eligible; those conditions should be assessed with the patient before registration in the trial
* Patients with major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after last dose
  Drug safety and tolerability will be evaluated by descriptively summarizing AEs, laboratory assessments, vital signs, and electrocardiogram assessments using tables of frequencies and counts for categorical variables and means (sds) or medians (ranges, interquartile ranges) for continuous variables.

SECONDARY OUTCOMES:
Overall survival | Up to 1 year
  The survival curve will be plotted using the Kaplan-Meier method. Median survival time and the 95% confidence interval will be presented for each study group and 1-year overall survival will be estimated. The 95% confidence intervals will be obtained by Greenwood?s formula.
Median survival | Up to 1 year
  The survival curve will be plotted using the Kaplan-Meier method. Median survival time and the 95% confidence interval will be presented for each study group and 1-year overall survival will be estimated. The 95% confidence intervals will be obtained by Greenwood?s formula.
Progression free survival at 6 months | Up to 6 months
  The Kaplan Meier curve will be plotted and median time to disease progression and the 95% confidence interval will be calculated. 6-month progression free survival will also be estimated. Since tumor assessment will only be performed periodically (every 8 weeks), the Kaplan-Meier estimate (estimated probability that a subject is progression-free at a specific time) and its 95% confidence interval will be provided at the end of each 8-week period.
Median time to disease progression | Up to 1 year
  The Kaplan Meier curve will be plotted and median time to disease progression and the 95% confidence interval will be calculated. 6-month progression free survival will also be estimated. Since tumor assessment will only be performed periodically (every 8 weeks), the Kaplan-Meier estimate (estimated probability that a subject is progression-free at a specific time) and its 95% confidence interval will be provided at the end of each 8-week period.
Radiographic response rates (RR) | Up to 3 years
  Response rate is the percentage of subjects who achieve partial response (PR) or complete response (CR) according to the immunotherapy Response Assessment in Neuro-Oncology (iRANO) criteria. Radiographic RR will be determined by iRANO criteria. The response rate will be calculated as the percentage of responders, and similarly, the 95% confidence interval will be calculated using the exact binomial method, if data allows.
Response rate | Up to 3 years
  Defined as percentage of subjects who achieve PR or CR according to the iRANO criteria. The response rate will be calculated as the percentage of responders, and similarly, the 95% confidence interval will be calculated using the exact binomial method, if data allows.
Median duration of response | Up to 1 year
  Tumor response will be reported as CR, PR, stable disease (SD), PD, or unknown according to the iRANO criteria. The response rate will be calculated as the percentage of responders, and similarly, the 95% confidence interval will be calculated using the exact binomial method, if data allows.

CONTACTS AND LOCATIONS:
Overall Officials: Rimas V Lukas, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Wainwright D, Lukas R, Zhai L, Lauing K, Kim M, Koch T, Penco-Campillo M, Bommi P, Dixit K, Kumthekar P, Sharp L, Lezon R, Garcia D, Sonabend A, McCortney K, Castro B, Chandler J, Gondi V, Grimm S, Heimberger A, Dobinda K, Zhang H, Sachdev S, Juhasz C, James CD, Allen J, Horbinski C, Lesniak M, Stupp R, Miska J. Newly diagnosed glioblastoma IDHwt patients treated with radiation, nivolumab, and BMS-986205. Res Sq [Preprint]. 2025 Sep 25:rs.3.rs-7567487. doi: 10.21203/rs.3.rs-7567487/v1. PMID 41041559

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT04047706/Prot_SAP_000.pdf